CLINICAL TRIAL: NCT06399731
Title: NEuroStimulation for the Treatment of Mild Cognitive Impairment in Parkinson's Disease: an Acceptability Cross-over Study
Brief Title: Non-invasive Brain Stimulation for the Treatment of Mild Cognitive Impairment in Parkinson's Disease
Acronym: NESCIO-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Tim Van Balkom, Post-doctoral researcher, Amsterdam UMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023.0804; 10390052210003 (Other Grant/Funding Number: ZonMw); NL84843.018.23 (Registry Identifier: ToetsingOnline)
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Four consecutive phases: 1) a no-intervention baseline phase, 2) rTMS or tDCS, 3) a second no-intervention baseline phase, 4) the second NIBS intervention. All phases have a duration of 4 weeks and the order of the NIBS interventions is counterbalanced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm 1: rTMS followed by tDCS (Experimental): Participants in intervention arm 1 will undergo four phases in the following order: 1) a no-intervention baseline phase, 2) 12 sessions of 20-minute institute-based repetitive transcranial magnetic stimulation (rTMS) (10 Hz) targeting the left DLPFC, 3) a second no-intervention baseline phase, 4) 20 sessions of 20-minute at-home anodal high-definition transcranial direct current stimulation (tDCS) targeting the left DLPFC. All phases have a duration of 4 weeks.
  Interventions: Device: High-frequency (10Hz) rTMS; Device: Anodal tDCS
- Intervention arm 2: tDCS followed by rTMS (Experimental): Participants in intervention arm 2 will undergo four phases in the following order: 1) a no-intervention baseline phase, 2) 20 sessions of 20-minute at-home anodal high-definition transcranial direct current stimulation (tDCS) targeting the left DLPFC, 3) a second no-intervention baseline phase, 4) 12 sessions of 20-minute institute-based repetitive transcranial magnetic stimulation (rTMS) (10 Hz) targeting the left DLPFC. All phases have a duration of 4 weeks.
  Interventions: Device: High-frequency (10Hz) rTMS; Device: Anodal tDCS

INTERVENTIONS:
Device: High-frequency (10Hz) rTMS — High-frequency (10 Hz) rTMS targeting the left DLPFC, based on fMRI-peak activation during performance of the Tower of London task, at 110% resting motor threshold intensity, corrected for scalp-cortex distance at the target location, for a total of 3000 pulses per session, using 30 trains of 10 seconds with 30-second inter-train intervals (total duration: 20 minutes), using neuronavigation to record the pulse location.
Device: Anodal tDCS — Anodal high-definition tDCS. The anode will be placed at the F3 EEG location, coordinates registered using neuronavigation on the first intervention session on-site, and cathodes at Fp1, Fz, C3 and F7, in a ring surrounding the anode, using π cm2 circular stimulation electrodes, stimulating the left DLPFC at 2 mA intensity for a duration of 20 minutes, 15 s ramp up and 15 s ramp down. After an initial on-site instructional tDCS session, the tDCS intervention will be delivered at home, in part remotely-supervised via MS Teams.

SUMMARY:
This cross-over pilot study aims to study the acceptability of two methods of non-invasive brain stimulation for the treatment of Parkinson's disease mild cognitive impairment (PD-MCI) - repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS) targeted at the left dorsolateral prefrontal cortex (DLPFC). Twenty participants will undergo both interventions in a cross-over design. They sequentially undergo four consecutive phases (4 weeks each), 1) no-intervention baseline, 2) rTMS ór tDCS, 3) no-intervention, 4) second intervention. The primary outcome measure will be acceptability of the interventions, and secondary outcomes include feasibility, cognitive function, neuropsychiatric symptoms, motor function. We will use MRI to explore personalized targeting.

DETAILED DESCRIPTION:
RATIONALE: Mild cognitive impairment (MCI) is a highly prevalent non-motor characteristic affecting about 40% of individuals with Parkinson's disease (PD). PD-MCI negatively impacts daily life functioning and quality of life and is associated with presence of other neuropsychiatric symptoms. Importantly, it constitutes a risk factor for later development of PD-related dementia.

Despite many endeavours to pharmacologically improve PD-MCI, there is currently no effective treatment. Optimization of dopaminergic therapy in early PD can relieve cognitive deficits, improving cognitive inflexibility and bradyphrenia, but also exacerbating other cognitive domains. Additionally, other non-pharmacological treatment options such as cognitive training have shown moderate effect sizes, but with limited transfer to daily functioning.

Non-invasive brain stimulation (NIBS) through repetitive transcranial magnetic stimulation (rTMS) or transcranial direct current stimulation (tDCS) has promise in treating PD-MCI. NIBS, particularly institute-based rTMS, is, however, intensive and complex in use, specifically for individuals with motor and cognitive difficulties, which might limit its potential for clinical use.

OBJECTIVE: To study the acceptability and feasibility of rTMS and tDCS for the treatment of individuals with PD-MCI.

STUDY DESIGN: A cross-over design with three conditions: a baseline condition, rTMS, and tDCS. The study consists of 1) two four-week intervention periods, with rTMS treatment three times a week (total session duration ~40 mins, treatment duration = 20 mins) and tDCS treatment five times a week (total session duration ~30 mins, treatment duration = 20 mins. For the rTMS intervention, stimulation will be performed at the Amsterdam UMC, location VUmc (and thus includes travel time); 2) one 120-minute assessment (baseline) that includes neuropsychological and motor assessment, and MR imaging, and four 60-minute assessments that only includes neuropsychological assessment.

STUDY POPULATION: We will enroll twenty individuals with PD-MCI, according to level I criteria by the Movement Disorders Society: Montreal Cognitive Assessment score range [21-25], performance 1-2 SD below appropriate norms on at least 2 neuropsychological tests, or recent (< 6 months) classification of PD-MCI on neuropsychological assessment elsewhere.

INTERVENTION: Participants will undergo four consecutive phases in this intervention study: 1) a no-intervention baseline phase, 2) 12 sessions of 20-minute institute-based repetitive transcranial magnetic stimulation (rTMS) (10 Hz) or 20 sessions of 20-minute at-home anodal high-definition transcranial direct current stimulation (tDCS) targeting the left dorsolateral prefrontal cortex (DLPFC), 3) a second no-intervention baseline phase, 4) the second alternative NIBS intervention. All phases have a duration of 4 weeks and the order of the NIBS interventions is counterbalanced.

MAIN STUDY PARAMETERS: The primary outcome measure will be acceptability of the interventions, and secondary outcomes include feasibility, cognitive function, neuropsychiatric symptoms, motor function. We will use MRI to explore personalized targeting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease, diagnosed by a neurologist;
* Mild to moderate disease stage (Hoehn & Yahr disease stage < 4);
* Movement Disorders Society level I criteria for PD-MCI (Litvan et al., 2012):

  * Montreal Cognitive Assessment score range [21-25] (Dalrymple-Alford et al., 2010), or
  * performance 1-2 SD below appropriate norms on at least 2 neuropsychological tests, or
  * classification of PD-MCI based on recent (< 6 months previous to participation) neuropsychological assessment taken elsewhere (report will be requested);- In case of (dopaminergic) medication use, participants are on stable medication for at least one month before participation and expect to remain on stable medication during the study

Exclusion Criteria:

* Indication for dementia based on the SAGE (cut-off ≤ 14; Scharre et al., 2010);
* Severe depressive disorder (Beck Depression Inventory - Ib score > 18);
* Psychotic disorder (except for benign hallucinations with insight), screened with the Scale for Assessment of Positive Symptoms for Parkinson's disease;
* Indication of alcohol or drug abuse;
* Contra-indication for rTMS according to Magstim Rapid2 Manual; rTMS should not be:

  * used on or in the vicinity of patients or users with cardiac demand pacemakers, implanted medication pumps, cochlear devices, implanted defibrillators and/or implanted neurostimulators
  * used on or in the vicinity of patients with implanted metal objects• used on patients where the skin in the area to be contacted is broken
  * used on those with large ischaemic scars
  * used on pregnant women
  * used on infants under the age of 2 years
  * used on epileptic individuals
  * used on those with a family history of convulsions
  * used on individuals with brain lesions that could affect seizure threshold
  * used on individuals suffering from multiple sclerosis
  * used on individuals taking tricyclic antidepressants, neuroleptic agents or any other drug that could lower seizure threshold,
  * used on individuals suffering from sleep deprivation during rTMS procedures
  * used on individuals with a heavy consumption of alcohol or those using epileptogenic drugs
  * used on individuals with severe heart disease or with increased intracranial pressure be used on those who have uncontrolled migraines
* Contra-indication for tDCS according to Neuroelectrics Starstim Manual; tDCS should not be used in case of:

  * Patients with a history of seizures;
  * Patients with unexplained episodes of loss of consciousness, since such condition could be related with brain alterations or epilepsy;
  * Patients with unstable or non-controlled neuropsychiatric illness;
  * Patients having implanted brain medical devices;
  * Patients with implanted pacemakers;
  * Patients having any electrically, magnetically or mechanically activated implant;
  * Patients having cardiac, neural or medication implants;
  * Patients having vascular clips or any other electrically sensitive support system in the brain;
  * Patients with serious brain injury;
  * Patients showing damage of skin at sites of stimulation (the device can only be used in healthy skin without wounds, otherwise the resistance to current can be altered);
  * Patients suffering from skin problems, such as dermatitis, psoriasis or eczema;
  * Patients suffering from severe or frequent headaches;
  * Patients with any serious life-threatening disease such as congestive heart failure, pulmonary obstructive chronic disease or active neoplasia;
  * Pregnant women (women of childbearing age should undertake a pregnancy test to confirm eligibility before treatment).
* Contra-indication for MR imaging:

  * metal in the body (pacemaker, port-a-cath, prosthesis, (cochlear) implant)
  * previous brain surgery
  * head trauma that resulted in unconsciousness for at least 1 hour
  * clips
  * (old metal containing) tattoo
  * irremovable piercings
  * irremovable metal braces
  * pregnancy
  * claustrophobia other problems lying still for 45 minutes
  * metal in the teeth
  * neurostimulator (including deep brain stimulation)
* Space-occupying lesion on MRI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Quantative acceptability of the interventions (measured seperately) | Eight weeks and sixteen weeks (after first and second intervention)
  Measured with Theoretical Framework of Acceptability questionnaire ("TFA-PD questionnaire") score, measuring seven domains of acceptability

SECONDARY OUTCOMES:
Qualitative acceptability assessment of both interventions | After study termination (i.e., all participants finished)
  Qualitative assessment from focus groups after study termination
Intervention compliance (feasibility) | Eight weeks and sixteen weeks (during first and second intervention)
  Percent of missed intervention sessions
Intervention attrition (feasibility) | After study termination (i.e., all participants finished)
  Count of dropped out participants
Usability of the tDCS device (feasibility) | Eight weeks or sixteen weeks (after tDCS intervention)
  System Usability Scale score
Subjective cognitive function | Four, eight, twelve and sixteen weeks
  PD-Cognitive Functional Rating Scale score
Subjective cognitive function | Four, eight, twelve and sixteen weeks
  Cognitive Failures Questionnaire score
Global cognitive function | Four, eight, twelve and sixteen weeks
  Montreal Cognitive Assessment score
Attention/mental processing speed | Four, eight, twelve and sixteen weeks
  Trail Making Test A time
Executive function | Four, eight, twelve and sixteen weeks
  Trail Making Test B time
Executive function/language | Four, eight, twelve and sixteen weeks
  Letter Fluency score
Executive function | Four, eight, twelve and sixteen weeks
  Tower of London Accuracy
Executive function | Four, eight, twelve and sixteen weeks
  Tower of London Reaction Time
Episodic Memory | Four, eight, twelve and sixteen weeks
  Rey Auditory Verbal Learning Test ("15 Woordentest") Direct Recall score
Episodic Memory | Four, eight, twelve and sixteen weeks
  Rey Auditory Verbal Learning Test ("15 Woordentest") Delayed Recall score
Episodic Memory | Four, eight, twelve and sixteen weeks
  Rey Auditory Verbal Learning Test ("15 Woordentest") Recognition score
Mental processing speed | Four, eight, twelve and sixteen weeks
  Symbol Digit Modalities Test score
Verbal attention | Four, eight, twelve and sixteen weeks
  Wechsler Adult Intelligence Scale IV-NL-Digit Span Forward
Working memory | Four, eight, twelve and sixteen weeks
  Wechsler Adult Intelligence Scale IV-NL-Digit Span Backwards/Sorting
Depressive symptoms | Four, eight, twelve and sixteen weeks
  Beck Depression Inventory-lb score
Anxiety symptoms | Four, eight, twelve and sixteen weeks
  Parkinson Anxiety Scale score
Functional mobility | Four, eight, twelve and sixteen weeks
  Timed Get-up and Go test score

OTHER OUTCOMES:
Structural and functional connectivity | Baseline
  Measured with MPRAGE, resting-state fMRI, task-based fMRI, DWI
Distance to optimal DLPFC stimulation target | Baseline
  Measured with optimal voxel coordinate based on task-based fMRI
Age | Baseline
Sex | Baseline
Education level | Baseline
  Years
Education level | Baseline
  Verhage score
Medication use | Baseline, four, eight, twelve and sixteen weeks
  Levodopa equivalent daily dosage
Disease duration | Baseline
  Years
Disease stage | Baseline
  Hoehn & Yahr stage
Motor symptom severity | Baseline
  MDS-Unified PD Rating Scale Motor Assessment motor score
Psychotic symptoms | Baseline
  Scale for the Assessment of Positive Symptoms for PD score
General cognitive function | Baseline
  Self-Administered Gerocognitive Exam
TMS adverse events | During rTMS intervention (week 4-8, or week 12-16)
  TMSens_Q adverse events questionnaire
tDCS adverse events | During tDCS intervention (week 4-8, or week 12-16)
  Adapted tDCS adverse events questionnaire
Visuospatial function | Baseline
  Benton Judgement of Line Orientation test score
Substance abuse | Baseline
  CAGE Adapted to Include Drugs
Intervention expectancy | Four weeks, eight weeks
  Credibility-expectancy questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will commit to adhere to the findability, accessibility, interoperability and re-usability (FAIR) of the data collected during this study by publishing and sharing coded data and analysis code on online repositories to the limits of Dutch GDP regulations.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Anonymized data will be made available after full data collection has finished, when first data cleaning has been performed and the primary endpoint analyses have been performed.
Access Criteria: A data sharing agreement or equivalent will be set up.